CLINICAL TRIAL: NCT06689982
Title: Tofacitinib in Patients With Amyotrophic Lateral Sclerosis: A Proof-of-concept Clinical Trials
Brief Title: Tofacitinib in Patients With Amyotrophic Lateral Sclerosis
Acronym: TALENT
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Turing-Darwin Laboratory; West Institute of Computing Technology, Chongqing, China (Unknown)
Responsible Party: Principal Investigator, yilong Wang, Vice President of Beijing Tiantan Hospital, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2024-144-02
Record Dates: First submitted 2024-07-22; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis; Clinical trial; Tofacitinib; Neuroinflammation
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neuroinflammatory Diseases | interventions — tofacitinib

STUDY DESIGN:
Intervention Model Description: tofacitinib (5mg per tablet)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tofacitinib (Experimental): This group will receive tofacitinib citrate sustained-release tablets at 180 consecutive days .
  Interventions: Drug: Tofacitinib tablets

INTERVENTIONS:
Drug: Tofacitinib tablets — All patients should be closely monitored for signs and symptoms of infection during and after treatment with tofacitinib tablets. If a patient develops a severe infection, opportunistic infection, or sepsis, medication should be discontinued. During treatment, patients with lymphocyte counts < 500 cells/mm^3 or ANC < 500 cells/mm^3 confirmed by repeated testing should be stopped. When 500≤ANC≤1000 cells/mm^3, administration should be interrupted, and if ANC returns to more than 1000 cells/mm^3, administration should be resumed. When hemoglobin < 8 g/dL or decreases by more than 2 g/dL, administration should be interrupted until hemoglobin values return to normal.

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a fatal neurodegenerative disease, of which motor-neuron's degeneration may be associated with neuroinflammation. Tofacitinib is a Janus kinase (JAK) inhibitor that affects cellular hematopoiesis and cellular immune function. At the same time, tofacitinib is suitable for rheumatoid arthritis, psoriatic arthritis, and ankylosing spondylitis. This study is a single center, single arm, proof of concept, clinical trial study, and it is planned to use tofacitinib to carry out a clinical trial to observe the treatment effect of ALS patients.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis is a fatal neurodegenerative disease characterized by progressive loss and dysfunction of upper and lower motor neurons located in the brain and spinal cord, further resulting in paralysis. In the occurrence and development of ALS, the degeneration of motor neurons may be related to neuroinflammatory response, often accompanied by excessive proliferation of microglia, astrocyte and oligodendrocyte. Tofacitinib is a Janus kinase (JAK) inhibitor. JAKs are intracellular enzymes that transport signals generated by cytokine or growth factor-receptor interactions on cell membranes, thereby influencing cellular hematopoietic processes and cellular immune function. At the same time, tofacitinib is a marketed drug suitable for rheumatoid arthritis, psoriatic arthritis, and ankylosing spondylitis. In this study, tofacitinib was selected to carry out a clinical randomized controlled trial to observe the treatment effect in ALS patients.

This study is a single center, single arm, proof of concept, clinical trial study. In this study, 12 patients will be enrolled. The treatment will be 1 tablet (5 mg) twice a day, and be administered continuously for a total of 180 days.

Follow up: Face to face interviews will be made on baseline, 30±3 days, 90±7 days, and 180±14 days.

The primary outcome measure was the difference of changes in ALSFRS-R scale scores at 30±3 days, 90±7 days, and 180±14 days from baseline.

Secondary outcomes included the incidence of invasive mechanical ventilation within 180 days , the changes in modified Norris scale scores, quality of life (ALSAQ-40, EQ-5D-5L), lung function, and electromyography indicators at 30±3 days, 90±7 days, and 180±14 days from baseline.

Exploratory outcomes included the changes in muscle strength, gait function, 7T-MRI imaging indicators, biomarkers in plasma and CSF, fatigue level, anxious level and depressive level, constipation clinical score, overactive bladder symptom score and CNS-BFS score at 30±3 days, 90±7 days, and 180±14 days from baseline; clinical progression within 180 days; the relationship between embryological etiology of ALS patients and the severity and progression in ALS patients, as well as the multiple group changes in ALS patients during disease progression.

Safe outcomes included the incidence in adverse event/severe adverse event, death, serious infection, malignant tumor, lymphoproliferative disease, major cardiovascular adverse events, thrombogenesis, abnormal lymphocytes and neutrophilic granuloaytopenia within 180 days.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old≤ age≤ 75 years old, males or females;
* Forced vital capacity ≥ 60% of predicted vital capacity during the screening period;
* The diagnosis conforms to the diagnostic criteria for amyotrophic lateral sclerosis on the Gold Coast;
* Based on the analysis of whether the subject significantly deviates from the baseline healthy elderly population, whole exome sequencing (WES) revealed that the embryonic lineage etiology was interpreted as CD8+ T lymphocyte group and Th1 highly activated, and patients with pathways related to neural repair and energy metabolism pathways that were not significantly inhibited;(1.Obtain genomic data of patient embryonic samples (blood or oral swab) through whole exome sequencing (WES) technology;2.Utilizing the Damage Assessment of Genome shotgun (DAGG) system developed by the Turing Darwin Laboratory team, rare coding mutations in patient genomic data are converted into an activity profile of signaling pathways (APSP). If the patient's embryonic genomic interpretation of APSP compared to the baseline healthy population's embryonic APSP shows high activation of CD8+ T lymphocyte group and Th1 activity, and non-significant inhibition of Treg, neural repair, and energy metabolism pathways, the patient may be included in the clinical trial;3.This step is analyzed by the Turing Darwin Laboratory team, and based on the entry criteria of the clinical trial (high activation of CD8+ T lymphocyte group and Th1 activity, and non-significant inhibition of Treg, neural repair, and energy metabolism pathways), a modeling setting for the APSP score threshold for ALS will be established. Patients above the threshold can be included in the trial.
* Subjects or their legal representatives clearly understand and voluntarily participate in the study and sign the informed consent form;
* Subjects (including male subjects) are willing to have no birth plan and voluntarily take effective contraceptive measures during the entire study period and within 3 months after the end of the study, and have no plan to donate sperm or eggs.

Exclusion Criteria:

* Patients who cannot cooperate with the clinical trial project cycle as determined by professional medical staff;
* Individual whose use of tofacitinib is forbidden;
* Absolute lymphocyte counts < 500 cells /mm^3, absolute neutrophil counts (ANC) < 1000 cells /mm^3 or hemoglobin level < 9 g/dL;
* Serious infection;
* Positive HIV test or history of positive test;
* Positive hepatitis C virus antibody or positive test history;
* Hepatitis B active infection (hepatitis B surface antigen positive and/or serum HBV DNA positive or serum HBV DNA > 2 × 10^8 IU/mL;
* Positive syphilis test result or positive test history;
* Lumbar spine diseases or malformation;
* Have other conditions known to be associated with motor neuron dysfunction that may confuse or obscure an ALS diagnosis;
* Other psychiatric disorders diagnosed according to DSM-V diagnostic criteria, or significant suicide intent;
* With severe hepatic insufficiency, renal insufficiency or severe cardiac insufficiency (severe hepatic insufficiency refers to ALT value≥2.0 times the upper limit of normal value or AST value≥2.0 times the upper limit of normal value; severe renal insufficiency refers to CRE≥1.5 times the upper limit of normal value or eGFR<40mL/min/1.73m^2; severe cardiac insufficiency refers to NYHA class 3-4);
* Permanently dependent on ventilator-assisted ventilation;
* Individual who have difficulty communicating verbally to the extent that they are unable to communicate, understand or follow instructions normally, and are unable to cooperate with treatment and evaluation;
* History of alcohol and drug abuse;
* Patients who are pregnant, breast-feeding, or who are likely to become pregnant and plan to become pregnant;
* Patients participating in other clinical trials or using other biological agents, drugs, or devices under investigation;
* Unable to be cooperative and complete the follow-up due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes of ALSFRS-R scale scores in ALS patients | day 180±14
  Amyotrophiclateral sclerosis functional rating scale revised(ALSFRS-R) is the most common evaluation indicator in ALS related research, with scores ranging from 0 to 48. The higher the score, the better the functional retention and the milder the symptoms.

SECONDARY OUTCOMES:
Incidence of invasive mechanical ventilation in ALS patients | 180 days
  The incidence of invasive mechanical ventilation in ALS patients.
Changes of modified Norris scale scores in ALS patients | day 30±3, 90±7, and 180±14
  The changes of modified Norris scale scores in ALS patients from baseline. The modified Norris scale is a self-assessment scale for ALS patients, with scores ranging from 0 to 120, with higher scores indicating better functional retention.
Changes of ALSAQ-40 scale scores in ALS patients | baseline, day 30±3, day 90±7, and day180±14
  The changes of ALSAQ-40 scale scores in ALS patients from baseline. The scale is an evaluation of the quality of life of ALS patients, with indicators including physical activity, dietary ability, social interaction ability, and emotional response. Simple and highly operable, it can be used for patients to self evaluate their quality of life, with scores ranging from 0 to 200. The higher the score, the milder the symptoms.
Changes in EQ-5D-5L scale scores in ALS patients | baseline, day 30±3, day 90±7, and day180±14
  The changes of EQ-5D-5L scale scores in ALS patients from baseline. It includes five dimensions(mobility, self-care, usual activities, pain/discomfort, anxiety/depression), and each dimension contains five levels of severity - no problem, minor problem, moderate problem, serious problem, extremely serious problem.
Changes of lung function in ALS patients | baseline, day 30±3, day 90±7, and day180±14
  The changes of lung function (forced vital capacity) in ALS patients from baseline. Value decline indicates worse outcome of ALS patients, or disease progression and disability.
Changes of electromyography indicators in ALS patients | baseline, day 30±3, day 90±7, and day180±14
  The changes of electromyography indicators in ALS patients from baseline. Muscle involvement will be assessed by needle electromyography, which analyzes muscle damage qualitatively based on spontaneous, motor unit action potential and recruitment. More muscle involvement indicates worse outcome of ALS patients, or disease progression and disability. The electromyographic indicators include the amplitude of CMAP, munix, and musix of different muscles.

OTHER OUTCOMES:
Changes of muscle strength in ALS patients | baseline, day 30±3, day 90±7, and day180±14
  The changes of muscle strength in ALS patients from baseline.
Changes of gait function in ALS patients | baseline, day 30±3, day 90±7, and day180±14
  The changes of gait function in ALS patients from baseline.
Changes of 7T MRI imaging indicators in ALS patients | baseline, day 30±3, day 90±7, and day180±14
  The changes of 7T MRI imaging indicators in ALS patients from baseline. 7T mainly observes the range and degree of iron deposition in the central anterior gyrus. 7T MRI enables the visualization and quantification of motor neuron degeneration in ALS patients, providing valuable information on the extent and distribution of neuronal loss in the brain and spinal cord.
Changes of biomarkers in plasma in ALS patients | baseline, day 30±3, day 90±7, and day180±14
  The changes of biomarkers in plasma in ALS patients from baseline, including neurofilament light chain protein (NFL), Janus kinase (JAK) enzymes (JAK1/JAK2, JAK1/JAK3, and JAK2/JAK3), signal transducers and activators of transcription (STAT), and phosphorylated STAT (p-STAT). They have the same units of measure.
Changes of biomarkers in CSF in ALS patients | day 180±14
  The changes of biomarkers in CSF in ALS patients from baseline, including neurofilament light chain protein (NFL), Janus kinase (JAK) enzymes (JAK1/JAK2, JAK1/JAK3, and JAK2/JAK3), signal transducers and activators of transcription (STAT), and phosphorylated STAT (p-STAT). They have the same units of measure.
Changes of fatigue level in ALS patients | baseline, day 30±3, day 90±7, and day180±14
  The changes of fatigue level (FSS scale scores) in ALS patients from baseline. FSS is a single dimensional fatigue scale with 9 items, requiring patients to rate the impact of fatigue on different functional areas on a 7-point scale, and then take the average score. The FSS score range is from 0 to 7, with higher scores indicating more fatigue.
Changes of anxious level in ALS patients | baseline, day 30±3, day 90±7, and day180±14
  The changes of anxious level (HAMA scale scores) in ALS patients from baseline. If the total score of HAMA exceeds 29 points, it may indicate severe anxiety. Exceeding 21 points indicates obvious anxiety. If it exceeds 14 points, there must be anxiety. Exceeding 7 points may indicate anxiety. If the score is less than 7, there are no anxiety symptoms.
Changes of depressive level in ALS patients | baseline, day 30±3, day 90±7, and day180±14
  The changes of depressive level (HAMD scale scores) in ALS patients from baseline. If the total score of HAMD exceeds 24 points, it may indicate severe depression. Exceeding 17 points may indicate mild or moderate depression. If it is less than 7 points, there are no depressive symptoms.
Changes of King's College Staging progression in ALS patients | 180 days
  Stage 1: This stage is characterized by symptoms limited to one region, such as muscle weakness or speech difficulties.
  Stage 2: Symptoms begin to spread to other regions, affecting more muscles and functions.
  Stage 3: Symptoms further progress, leading to significant disability but with some independence in daily activities.
  Stage 4: Severe disability where the individual requires assistance for most activities of daily living.
  Stage 5: Advanced stage with total dependence on others for care and assistance.
Changes of MiToS Staging progression in ALS patients | 180 days
  Stage 1: Early stage with symptoms limited to one region or limb. Stage 2: Symptoms spread to other regions or limbs. Stage 3: Symptoms progress to involve both upper and lower limbs. Stage 4: Respiratory muscles become affected, leading to breathing difficulties.
  Stage 5: Severe respiratory impairment requiring ventilation support.
Correlation between germline etiology and ALS disease progression | 180 days
  The severity and progression rate of the disease will be assessed before enrollment into the clinical trial. After enrollment, blood will be drawn for whole exome sequencing. Through the newly developed multilevel data-driven AI modelDamage Assessment of Genomic shotGun(DAGG) by TD-LAB, the rare coding variations (gRCVs) in the germ line genome will be translated into functional spectra of hundreds of cellular functions and signaling pathways (including growth factors, immune functions, nerve repair, and other related functional pathways) to identify potential pathogenic factors in ALS patients. Furthermore, in conjunction with the patient's clinical phenotype, the correlation between the severity of the pathogenicity encoded by the germ line genome and the progression of ALS disease will be determined. And the disease progression of the disease will be comprehensively evaluated through electromyography, the ALSFRS-R scale, lung function tests, and physical examinations.
The Wexner Constipation Score in ALS patients | baseline, day 30±3, day 90±7, and day180±14
  The changes of constipation clinical score in ALS patients from baseline. This scoring system consists of several questions related to bowel habits, such as frequency of bowel movements, difficulty in passing stool, feeling of incomplete evacuation, and use of laxatives. Each question is assigned a score based on the severity of the symptom, with higher scores indicating more severe constipation. The score is ranging from 0 to 30.
Overactive Bladder Syndrome Score (OABSS) Overactive Bladder Syndrome Score (OABSS) Overactive Bladder Syndrome Score (OABSS) Overactive Bladder Syndrome Score (OABSS) in ALS patients | baseline, day 30±3, day 90±7, and day180±14
  The changes of OABSS in ALS patients from baseline. Change in Overactive Bladder Syndrome Score (OABSS, from 0 to 15, score increase indicates worse outcome of ALS patients, or disease progression and disability).
CNS-BFS score in ALS patients | baseline, day 30±3, day 90±7, and day180±14
  The changes of CNS-BFS score in ALS patients from baseline.
Multiple Omics Changes in ALS Patients During IIT Treatment | baseline, day 30±3, day 90±7, and day180±14
  This study will assess the multi-omics changes (including genomics, transcriptomics, and proteomics data) in ALS patients during the treatment process, analyze the correlation between multi-omics data and clinical manifestations, and drug responses to evaluate the multi-omics changes as the condition of ALS patients changes.
Security purpose：adverse event | day180±14
  The number of adverse event within 180 days. Adverse medical events occurring in subjects during the use of the investigational drug, or worsening of pre-existing medical conditions, regardless of causality with the investigational drug treatment, should be reported. Adverse medical events can be clinical symptoms/signs, diseases, or abnormal test results. Adverse events (AEs) encompass any adverse medical events that occur at any time during the entire clinical study, including the screening or washout periods, even if the patient has not yet received the investigational drug treatment.
Security purpose：severe adverse event | day180±14
  The number of evere adverse event within 180 days. Adverse events meeting one or more of the following criteria during the study period:
  * Result in death
  * Pose an immediate life-threatening condition Note: Life-threatening is defined as an event that at the time of occurrence places the patient in immediate danger of death, not necessarily an event that would have caused death if it were more severe.
  * Require hospitalization or prolongation of existing hospitalization
  * Result in persistent or significant disability/incapacity, or loss of a major ability to maintain normal life functions
  * Congenital anomaly, congenital defect, birth defect, or fertility impairment
  * Significant medical events that may jeopardize the subject or require medical intervention to prevent the above outcomes.
Security purpose：serious infection | day180±14
  The number of serious infection within 180 days. This refers to severe infections that have spread throughout the body, not just in one small area, which can be potentially life-threatening, requiring urgent medical attention and often hospitalization.
Security purpose：malignant tumor | day180±14
  The number of malignant tumor within 180 days. malignant tumor refers to a mass or growth of abnormal cells that are cancerous and can spread to other parts of the body or invade surrounding tissues, causing serious health problems.
Security purpose：lymphoproliferative disease | day180±14
  The number of lymphoproliferative disease within 180 days. This is a type of disease where lymphocytes, a type of white blood cell, are produced in excessive quantities. This may lead to immune system dysfunction and increase the risk of infections or cancer.
major cardiovascular adverse events | day180±14
  The number of major cardiovascular adverse events within 180 days. It refers to serious, unwanted health occurrences related to the cardiovascular system like heart attacks, strokes, heart failures or death.
Security purpose：thrombogenesis | day180±14
  The number of thrombogenesis within 180 days. The process of clot formation within blood vessels, which can block the flow of blood, leading to serious conditions such as stroke or heart attack.
Security purpose：abnormal lymphocytes | day180±14
  The number of abnormal lymphocytes within 180 days. Abnormal lymphocytes are lymphocytes, a type of white blood cell, that appear abnormal under a microscope. They may be unusually large or small, or have an unusual shape or structure, which could be a sign of an infection or disease like leukemia.
Security purpose：neutrophilic granuloaytopenia | day180±14
  The number of neutrophilic granuloaytopenia within 180 days. This is a condition characterized by a low level of neutrophils, a type of white blood cell important for fighting off infections, particularly those caused by bacteria and fungi. When the neutrophil count is low, it makes a person more vulnerable to infectious diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wang, PhD+MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No